| INFORMED CONSENT FORM FOR PARTICIPATION IN THE STUDY | |
|---|---|
| Study Title: | ROLE OF VERY LOW-CALORIE KETOGENIC DIET (VLCKD) IN PATIENTS WITH NON-ALCOHOLIC STEATOHEPATITIS (NASH) WITH FIBROSIS |
| Study Code: | KETONASH |
| Sponsor: | Department of Medical and Surgical Sciences (DIMEC) - Alma Mater Studiorum – University of Bologna |
| Principal<br>Investigator: | Prof. Fabio Piscaglia, Internal Medicine, Hepatobiliary, and Immunology Allergology Unit |
| Collaborators: | Dr. Federico Ravaioli, Prof. Maria Letizia Petroni, Dr. Silvia Garelli, Dr. Federica Perazza, Dr. Eleonora Terzi, Dr. Silvia Ferri, Dr. Simona Leoni, Dr. Francesco Tovoli, Prof. Alessandro Granito. |

## Dear Sir/Madam,

We intend to conduct medical-scientific research on this site, specifically an interventional study without devices and medications.

This study aims to evaluate, in patients with metabolic-associated fatty liver disease (MAFLD) with non-alcoholic steatohepatitis (NASH) and significant liver fibrosis, the effect of a very-low-calorie ketogenic diet (VLCKD) compared to a standard low-calorie diet (standard Mediterranean LCD - following the European EASL/ESPEN nutritional guidelines on MAFLD/NAFLD).

Participation in a study is an important decision. Before you decide to accept or refuse to participate, we ask you to read this information sheet carefully, taking all the time you need. You must seek clarification if anything is unclear or need further information. Additionally, if you wish, you can seek the opinion of your family members or a trusted medical professional before deciding. If you choose not to participate in the study, you will still receive all the therapies prescribed for your condition, and the doctors and other healthcare professionals will continue to follow you with due attention. Your decision to refrain from participating will not be interpreted as a lack of trust in their abilities.

### Why are we proposing your participation in this study?

We are inviting you to participate in this study because you are being treated at the Internal Medicine, Hepatobiliary, and Immunology Allergology Unit and have non-alcoholic steatohepatitis (NASH) with fibrosis, along with obesity.

### What does this study propose?

We have decided to conduct this study to assess the effect of a very low-calorie ketogenic diet (VLCKD) compared to a standard low-calorie diet (standard Mediterranean LCD).

The primary objective of the study is to evaluate MAFLD/NAFLD patients treated with VLCKD compared to standard LCD in the

- 1. Improvement in terms of liver fibrosis without worsening of NASH
- 2. Improvement in NASH without worsening of liver fibrosis

What does participation in this study entail compared to standard care, and what are your responsibilities as a participant?

#### **KETONASH**

Participation in the study involves a 6-month dietary intervention phase (Visits 1-8), followed by a 6-month weight maintenance phase (Visits 9-14). In both study arms, the intervention will be carried out using a standardised multidisciplinary approach (Physician/Dietitian/Nurse/Psychologist) aimed at weight loss through changes in diet, exercise, and emotional support techniques. The two study arms differ in nutritional composition, food types, and caloric intake. Participation in the study is free of charge and will not be rewarded in any way.

# What are the risks or inconveniences of participating in this study?

Participation in the study does not involve additional risks, except for the risks associated with executing the end-of-study liver biopsy, similar to the procedure performed in routine clinical practice. These risks may include bleeding, pain, visceral perforation, and blood pressure drop. Additionally, side effects related to the ketogenic diet may occur, such as headache, constipation, vitamin deficiencies, mineral deficiencies, nausea, vomiting, fatigue, and halitosis.

# What are the possible benefits of participating in this study?

Participating in the study will allow you to undergo an innovative dietary regimen under strict medical supervision, with in-depth monitoring for non-alcoholic steatohepatitis.

# Can you choose not to participate or change your mind?

Participation in this study is voluntary. You can refuse to participate or withdraw from the study at any time without giving any explanation and without any penalty or negative consequences. Your refusal to participate or the decision to discontinue participation will not affect the care you receive, which will still be the best available.

Any new information that may affect your decision to continue or discontinue participation in the study will be communicated to you as soon as possible. The same applies to any potential termination or suspension of the study.

### Do you need to inform your treating physician?

Considering the study design, if you decide to participate, it is essential to inform your general practitioner. We have prepared (or will provide you with) a letter explaining the study procedures to facilitate this.

#### **Insurance Coverage**

Please be informed that a specific insurance policy has been taken to cover any risks associated with your participation in this study. The insurance company is Lloyd's Insurance Company S.A., Policy Number: A1202150832-LB—coverage per participant: Euro 1,500,000.00; aggregate coverage: Euro 3,000,000.00. If you wish to claim compensation for damages due to participation in this study, you must request it within 24 months from the end of the study. If desired, you will receive a copy of the insurance terms and conditions at the time of consent signing.

#### **Access to Original Medical Documentation**

Direct access to your original medical documentation will be granted to those involved in monitoring or verification, the Ethics Committee, and regulatory authorities to verify study procedures and/or data without violating your confidentiality, to the extent permitted by applicable laws and regulations. By signing the informed consent form, you are authorising such access. Documents identifying you will be kept confidential and, to the extent permitted by laws and/or applicable regulations, will not be publicly available.

Regarding the treatment of your data, please read the information document.

## Has this study been approved by institutional bodies?

The study has been approved by the Independent Ethics Committee of the Emilia Centro Wide Area (CE-AVEC) of the Emilia-Romagna Region. The Ethics Committee is an independent body composed of internal and external members responsible for providing public assurance of the protection of rights, safety, and well-being of subjects participating in a clinical trial, expressing an opinion on ethics and scientificity before the start of any study involving humans.

# Information about Study Results

If interested and upon request, you will be informed of the general results of the study at the end of the experimentation. The results of this study may be presented at conferences or published; in any case, your name and other personal data that can identify you will not be included in any presentation or publication.

The protocol of this study and this information sheet have been prepared in accordance with Good Clinical Practice and the Declaration of Helsinki and have been approved by the Ethics Committee of the Emilia Centro Wide Area (CE-AVEC).

# Who can be contacted for any clarification about the study?

You can contact the Study Coordinator, the head of the centre you have approached, Prof. Fabio Piscaglia, at the following contact details:

Prof. Fabio Piscaglia

Internal Medicine, Hepatobiliary, and Immunology Allergology Unit Via Albertoni 15, Bologna, Italy Tel: 0512142214 Email: fabio.piscaglia@unibo.it

Thank you for your attention, for considering the possibility of participating in the study, and for the time dedicated to reading this information sheet. Please keep this document

and bring it if you decide to participate in the study.

| INFO | RMED CONSENT FORM FOR PARTICIPATION IN THE STUDY |
|---|---|
| Study Title: | ROLE OF VERY LOW-CALORIE KETOGENIC DIET (VLCKD) IN PATIENTS WITH NON-ALCOHOLIC STEATOHEPATITIS (NASH) WITH FIBROSIS |
| Study Code: | KETONASH |
| Sponsor: | Department of Medical and Surgical Sciences (DIMEC). Alma Mater<br>Studiorum – University of Bologna |
| Principal<br>Investigator: | Prof. Fabio Piscaglia, Internal Medicine, Hepatobiliary, and Immunology<br>Allergology Unit |
| Collaborators: | Dr. Federico Ravaioli, Prof. Maria Letizia Petroni, Dr. Silvia Garelli, Dr. Laura Leoni, Dr. Federica Perazza, Dr. Eleonora Terzi, Dr. Silvia Ferri, Dr. Simona Leoni, Dr. Francesco Tovoli, Prof. Alessandro Granito. |
| Place of Birth: Residing at: Email: Phone: | d: |
| in the stu - To have r - To have r - To under without p - Be awar collected | received comprehensive explanations regarding the request to participate dy, mainly its purposes and procedures. nad the opportunity to ask questions and receive satisfactory answers. read and understood the information sheet provided well in advance. restand that participation is voluntary, they can withdraw from the study roviding explanations, which will not affect their future care. re that if they withdraw their consent, the researcher will use the data before consent withdrawal. responsibility for delivering the letter regarding the study to their general er. |
| - Freely accepts | vith these statements:<br>s to participate in the study.<br>ontacted in the future to provide new information. |
| | Signature: |
| | ame:Signature: |
| • | al Witness (if necessary): |
| _ | Signature: |

# NOTES:

1 copy for the Patient, 1 copy for the Investigator, and 1 copy to be retained in the Patient's medical record.